CLINICAL TRIAL: NCT07146789
Title: Effectiveness of the Home-Based Graded Repetitive Arm Supplementary Program Combined With Occupational Therapy Versus Conventional Occupational Therapy Alone on Quality of Life and Upper Limb Function After Stroke: A Randomized Controlled Trial
Brief Title: Home-based Graded Repetitive Arm Supplementary Program for Quality of Life and Functional Upper Limb Recovery
Acronym: REC-HOMEGRASP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Hermanas Hospitalarias del Sagrado Corazón de Jesús, Spain (Unknown)
Responsible Party: Principal Investigator, Eva María Navarrete Muñoz, Doctora por la Universidad Miguel Hernandez de Elche, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 240408194759
Record Dates: First submitted 2025-07-31; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Stroke With Hemiparesis
Keywords: stroke; hemiparesis; upper limb; upper extremity; recovery
MeSH Terms: conditions — Stroke; Paresis | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: This is a single-blind, two-arm, parallel-group, randomised controlled trial to evaluate the effectiveness of the Spanish version of the HomeGRASP programme as an adjunct to conventional occupational therapy in adults post-stroke. Participants will be randomly assigned to: (1) Control group: conventional occupational therapy (2-3 sessions/week, 45 minutes each) including task-oriented training, ADL training, and mobilisation if needed (max. 10 min); or (2) Intervention group: the same conventional therapy plus the HomeGRASP programme (1 hour/day, 7 days/week for 8 weeks), supervised weekly by an occupational therapist, who reviews and adjusts the exercise plan during the session. Assessments will be performed at baseline and post-intervention by a blinded evaluator.
Who Masked: Outcomes Assessor
Masking Description: The principal investigator will carry out the statistical analysis without any contact with the participants or involvement in data collection. All participant assessments will be conducted by an external evaluator who is not involved in the implementation of the intervention or the project team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HomeGRASP and occupational therapy (Experimental): The experimental group will carry out the conventional treatment described in the control group together with the HomeGRASP programme at home. This programme consists of one hour of exercises at home, seven days a week, for a period of eight weeks. As the programme involves supervision by the occupational therapist of the exercises carried out at home, 20-30 minutes of the conventional session will be devoted to reviewing this plan. Before the programme starts, an explanatory session will be held with the patient and, if necessary, with the carer to show and teach the correct way to do the exercises proposed in the programme, as well as providing the material needed to do them.
  Interventions: Other: occupational therapy combined with HomeGRASP program
- Grupo control (Active Comparator): The control group will only receive conventional occupational therapy treatment at the rehabilitation centre. The conventional treatment sessions will be based on: generally between 2-3 sessions a week lasting 45 minutes each at the rehabilitation centre they attend. The approaches that will be used during the sessions will be based solely on mobilisations of the affected upper limb if necessary (maximum 10 minutes of the session), task-oriented training and training in ADLs.
  Interventions: Other: occupational therapy

INTERVENTIONS:
Other: occupational therapy combined with HomeGRASP program — To the present date there has been no trial combining conventional treatment with the GRASP programme as opposed to conventional treatment alone. Therefore, it is necessary to translate and adapt the materials transculturally so that it can be applied in Spain and verify the changes that occur in perceived quality of life and functionality of the affected upper limb as primary outcomes, as well as evaluating manipulative skills, use of the upper limb in ADLs and personal autonomy as secondary outcomes. All this, through the HomeGRASP programme as a complement to conventional rehabilitation in occupational therapy.
  Arms: HomeGRASP and occupational therapy
Other: occupational therapy — It will consist solely of conventional occupational therapy treatment at the rehabilitation centre. The conventional treatment sessions will be based on: generally between 2-3 sessions a week lasting 45 minutes each at the rehabilitation centre you attend. The approaches to be used during the sessions will be based solely on mobilisations of the affected upper limb if necessary (maximum 10 minutes of the session), task-oriented training and training in ADLs.
  Arms: Grupo control

SUMMARY:
In post-stroke rehabilitation of the affected upper limb, increasing treatment intensity has been shown to lead to better outcomes compared to conventional approaches with fewer hours of therapy per day and week. However, logistical, human, and material constraints in neurorehabilitation centres often limit the feasibility of increasing treatment intensity.

The GRASP programme (Graded Repetitive Arm Supplementary Program) is a home-based exercise intervention grounded in motor learning principles and conducted weekly under the supervision of an occupational therapist. This strategy enables the intensity of upper limb rehabilitation to be increased by up to seven additional hours per week.

This project aims to evaluate the effectiveness of the Spanish version of the HomeGRASP programme, implemented as an adjunct to conventional occupational therapy, in improving quality of life, autonomy, and upper limb functionality in people after stroke. To this end, a single-blind, randomised controlled clinical trial will be conducted. Participants in the experimental group will receive conventional occupational therapy in addition to the HomeGRASP programme performed at home, while those in the control group will receive only conventional therapy. The treatment period for both groups will last eight weeks.

Participants will be assessed at baseline and after the 8-week intervention period by a blinded evaluator. The primary outcomes will include changes in quality of life and upper limb functionality, measured using the CAVIDACE scale and the Wolf Motor Function Test. Secondary outcomes will include upper limb dexterity and personal autonomy, assessed using the Box and Block Test, Purdue Pegboard Test, Motor Activity Log-30, Duruöz Hand Index, and the Functional Independence Measure (FIM).

DETAILED DESCRIPTION:
Stroke is a sudden neurological event that can cause temporary or permanent impairments depending on the brain area affected. Among the resulting deficits, the loss of upper limb functionality on the affected side is one of the greatest challenges in rehabilitation. It is estimated that at least 80% of stroke survivors experience some degree of upper limb dysfunction, while only about 15% achieve significant functional recovery. Given the critical role of the arms and hands in performing activities of daily living (ADLs), such impairments can severely reduce a person's independence and contribute to long-term disability.

Recent studies have highlighted that the time allocated for upper limb rehabilitation in standard care is often insufficient. Increasing the intensity of therapy has been shown to yield better functional outcomes, especially in the chronic phase of stroke recovery. Strategies to increase intensity include extending the duration of therapy sessions and promoting a higher number of task repetitions, which support motor learning and functional generalisation. While technologies such as robotics and virtual reality are being used to deliver more intensive therapy at home, they often come with increased costs and usability barriers, particularly for older adults or those unfamiliar with digital tools.

A practical solution is the implementation of structured home-based exercise programmes. One such programme is the Graded Repetitive Arm Supplementary Program (GRASP), developed by the University of British Columbia. GRASP consists of a set of 33 structured exercises targeting various aspects of upper limb rehabilitation, including stretching, strength, coordination, and fine motor skills. It is delivered in a self-directed format with weekly supervision by an occupational therapist. The programme includes initial in-person instruction, delivery of all required materials, and weekly monitoring through exercise logs and patient feedback. Pain levels are tracked using a visual analogue scale to ensure patient safety and guide therapy adjustments. The standard application involves performing one hour of daily exercises, seven days a week, over an eight-week period.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age.
* Have suffered only one stroke and be clinically stable.
* At least 3 months must have passed since the stroke and less than 12 months.
* Signing of informed consent
* Be able to communicate any adverse effects (e.g. shoulder pain)
* Be able to follow instructions and perform the exercises independently for one hour. If they are not able to do so, have the help of a caregiver to ensure that the exercises are performed.
* Perform at least 10º of active wrist or finger extension.
* Ability to raise the scapula of the affected upper limb against gravity.

Exclusion Criteria:

* Having neurological conditions other than stroke.
* Experiencing excessive pain in the affected upper limb that prevents the patient from correctly performing the exercises proposed in the programme. Visual Analogue Scale (VAS > 7).
* Having a visual perception deficit that prevents the patient from correctly performing the exercises proposed in the programme.
* Excessive muscle tone (spasticity or hypertonia) that prevents the person from correctly performing the exercises proposed in the programme. Asworth > 2.
* A Folstein Mini-Mental State Examination (MMSE) score of ≥22 is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Functionality of the affected upper limb through tasks | 2 month
  Wolf Motor Function Test (WMFT): quantifies the motor capacity of the upper limbs (UL) through timed and functional tasks. The tool consists of 17 elements including 6 items involving timed functional tasks, items 7 and 14 are measures of strength, and the remaining 9 items consist of analysing the quality of movement when completing various tasks.
Quality of life as perceived by the patient | 2 months
  CAVIDACE: this is an evaluation of the perceived quality of life of adults with brain damage from the perspective of an external evaluator. It is recorded by a person who knows the user well (e.g. professionals, family members, legal guardians...). The sections included in this tool are: emotional well-being, interpersonal relationships, material well-being, personal development, physical well-being, self-determination, social inclusion and rights.

SECONDARY OUTCOMES:
Assess the gross motor skills of the patient's affected upper limb | 2 months
  Box and Blocks Test (BBT): this is an assessment tool that measures a person's gross unimanual motor skills. It consists of moving the maximum number of wooden blocks from one side of the box to the other in one minute.
Assessing the fine motor skills of the patient's affected upper limb | 2 months
  Purdue Pegboard Test (PPT): this test aims to measure the unimanual and bimanual dexterity of the fingers, the gross movement of the hands and arms in patients with upper limb deficiencies as a result of neurological and musculoskeletal conditions. It consists of a board with two parallel rows with 25 holes in which different metal pegs, washers and tubes are placed, which are located in the upper part of the board in four cavities. It has four parts: the first assesses the dexterity of the dominant hand, the second the non-dominant hand, the third evaluates simultaneous bimanual coordination and the last measures alternating bimanual coordination through an assembly task.
To assess the real use of the affected upper limb in activities of daily living. | 2 months
  Motor Activity Log-30 (MAL): this consists of a questionnaire with 30 items in which the amount and quality of use of the upper limb affected after a stroke is subjectively assessed when carrying out different tasks of daily living. The score for each item varies between 0 (does not use the affected arm to carry out the activity) and 5 (includes the affected hand in the same way as before the stroke).
Assessing the difficulty patients have when carrying out daily activities with their hands. | 2 months
  The Duruöz Index (DI), also called the Cochin Scale, contains 18 questions and is a self-administered scale that measures the difficulty of performing ADLs such as cooking, dressing, personal hygiene, office tasks, etc. Patients rate their ability from 0 (no difficulty) to 5 (impossible to perform).
Valuing the independence of the patient in activities of daily living. | 2 months
  Functional Independence Measure (FIM): this is an 18-item global measure of disability. Each item has seven ordinal levels of scoring from 1 (total care) to 7 (total independence) in order to quantify the functional independence of the person being evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Soler Pons, Occupational Therapy, Study Director — Fundación Hospitalarias Valencia; Eva María Navarrete Muñoz, Phd, Principal Investigator — Universidad Miguel Hernández de Elche; Desirée Valera Gran, Phd, Principal Investigator — Universidad Miguel Hernández de Elche
Locations (1):
- Fundación Hopitalarias, Centro sociosanitario Nuestra señora del Carmen, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang CL, Waterson S, Eng JJ. Implementation and Evaluation of the Virtual Graded Repetitive Arm Supplementary Program (GRASP) for Individuals With Stroke During the COVID-19 Pandemic and Beyond. Phys Ther. 2021 Jun 1;101(6):pzab083. doi: 10.1093/ptj/pzab083. PMID 33682872
- [Background] Simpson LA, Eng JJ, Chan M. H-GRASP: the feasibility of an upper limb home exercise program monitored by phone for individuals post stroke. Disabil Rehabil. 2017 May;39(9):874-882. doi: 10.3109/09638288.2016.1162853. Epub 2016 Mar 26. PMID 27017890
- [Background] Connell LA, McMahon NE, Watkins CL, Eng JJ. Therapists' use of the Graded Repetitive Arm Supplementary Program (GRASP) intervention: a practice implementation survey study. Phys Ther. 2014 May;94(5):632-43. doi: 10.2522/ptj.20130240. Epub 2014 Feb 6. PMID 24505098
- [Background] Connell LA, McMahon NE, Harris JE, Watkins CL, Eng JJ. A formative evaluation of the implementation of an upper limb stroke rehabilitation intervention in clinical practice: a qualitative interview study. Implement Sci. 2014 Aug 12;9:90. doi: 10.1186/s13012-014-0090-3. PMID 25112430
- [Background] Harris JE, Eng JJ, Miller WC, Dawson AS. A self-administered Graded Repetitive Arm Supplementary Program (GRASP) improves arm function during inpatient stroke rehabilitation: a multi-site randomized controlled trial. Stroke. 2009 Jun;40(6):2123-8. doi: 10.1161/STROKEAHA.108.544585. Epub 2009 Apr 9. PMID 19359633
- [Background] Essers B, Veerbeek JM, Luft AR, Verheyden G. The feasibility of the adapted H-GRASP program for perceived and actual daily-life upper limb activity in the chronic phase post-stroke. Disabil Rehabil. 2024 Dec;46(24):5815-5828. doi: 10.1080/09638288.2024.2313121. Epub 2024 Feb 8. PMID 38329448
- See also: Web page about original GRASP program — https://neurorehab.med.ubc.ca/grasp/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT07146789/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT07146789/ICF_001.pdf